CLINICAL TRIAL: NCT05264493
Title: A PHASE 1 RANDOMIZED, OPEN-LABEL, SINGLE-DOSE, 3-TREATMENT CROSS-OVER STUDY TO EVALUATE RELATIVE BIOAVAILABILITY OF INTRAMUSCULAR INJECTION OF NALOXONE HCL 5 Milligrams (mg) [5mg/0.5 Milliliters (mL] USING A QUICKSHOT™ AUTOINJECTOR COMPARED TO 2 mg NALOXONE INTRAMUSCULAR INJECTION AND 2 mg NALOXONE INTRAVENOUS INJECTION IN HEALTHY ADULT PARTICIPANTS
Brief Title: Bioavailability Study of Naloxone 5 Milligrams (mg) Intramuscular (IM) Autoinjector
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: C2431001
Record Dates: First submitted 2022-02-14; First posted 2022-03-03 (Actual); Last update posted 2022-03-03 (Actual); Status verified 2022-03

CONDITIONS: Healthy Volunteers
Keywords: naloxone; autoinjector; intramuscular; high dose; 5 mg; healthy volunteers; safety; cross-over study; pharmacokinetics; 3 treatment arms
MeSH Terms: interventions — Naloxone

STUDY DESIGN:
Intervention Model Description: Williams Square Study Design with 6 sequences
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- naloxone 5 mg IM autoinjector (Experimental): participants will receive in random order, a single naloxone 5 mg IM autoinjector injection into the lateral thigh
  Interventions: Drug: NaxRedy ™
- naloxone 2 mg IM (Active Comparator): participants will receive in random order, a single naloxone 2 mg IM injection into the gluteus muscle
  Interventions: Drug: Naloxone Hydrochloride Injection, USP
- naloxone 2mg bolus IV (Active Comparator): participants will receive in random order, a single naloxone 2 mg bolus IV injection
  Interventions: Drug: Naloxone Hydrochloride Injection, USP

INTERVENTIONS:
Drug: NaxRedy ™ — 5 mg (5 mg/0.5 mL) IM autoinjector injection into lateral thigh
  Arms: naloxone 5 mg IM autoinjector
Drug: Naloxone Hydrochloride Injection, USP — 2 mg IM (2mg/2 mL) injection into gluteal muscle
  Arms: naloxone 2 mg IM
Drug: Naloxone Hydrochloride Injection, USP — 2 mg bolus IV (2mg/2 mL)
  Arms: naloxone 2mg bolus IV

SUMMARY:
To compare the plasma concentration (bioavailability) and safety of a single naloxone 5 mg autoinjector intramuscular (IM) injection to a single 2 mg IM injection (an approved safe dose) and to a single 2 mg bolus intravenous (IV) injection (an approved safe dose)

DETAILED DESCRIPTION:
A randomized, open-label, 3-treatment, 6-sequences, 3-period Williams Square crossover single-dose, relative bioavailability study in healthy adult participants. The study includes Screening period, a Treatment period and a Follow-up contact (SoA). At least twelve (12) participants will be enrolled. If the number of evaluable participants falls below 12, participants may be replaced.

ELIGIBILITY:
Inclusion Criteria:

Participants are eligible to be included in the study only if all of the following criteria apply:

Age and Sex:

1. Healthy male and/or female participants of non-childbearing potential, who, at the time of screening, are between the ages of 18 and 55 years, inclusive.

   Refer to protocol for reproductive criteria for male and female participants.

   Type of Participant and Disease Characteristics:
2. Male and female participants who are overtly healthy as determined by medical evaluation including medical history, physical examination, vital signs, 12-lead ECG, and/or clinical laboratory tests.
3. Participants who are willing and able to comply with all scheduled visits, treatment plan, laboratory tests, lifestyle considerations, and other study procedures.

   Weight:
4. BMI of 17.5 to 30.5 kg/m2; and a total body weight > 50 kg (110 lb).

Informed Consent:

5. Capable of giving signed informed consent as described in Appendix 1, which includes compliance with the requirements and restrictions listed in the ICD and in this protocol.

-

Exclusion Criteria:

Participants are excluded from the study if any of the following criteria apply:

Medical Conditions:

1. Other medical or psychiatric condition including recent (within the past year) or active suicidal ideation/behavior or laboratory abnormality that may increase the risk of study participation or, in the investigator's judgment, make the participant inappropriate for the study.
2. Current or past diagnosis of any type of drug dependence within the past year will not be eligible to participate. History of alcohol abuse, dependence or binge drinking and/or any other illicit drug use within 6 months of screening. Binge drinking is hours. As a general rule, alcohol intake should not exceed 14 units per week (1 unit = 8 ounces (240 mL) beer, 1 ounce (30 mL) of 40% spirit or 3 ounces (90 mL) of wine).
3. If fever is present within 7 days of admission or screening.
4. Evidence or history of clinically significant hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, neurological, or allergic disease (including drug allergies, but excluding untreated, asymptomatic, seasonal allergies at the time of dosing).
5. History of HIV infection, hepatitis B, or hepatitis C, positive testing for HIV, HBsAg, or HCVAb. Hepatitis B vaccination is allowed.
6. Other medical or psychiatric condition including recent (within the past year) or active suicidal ideation/behavior or laboratory abnormality that may increase the risk of study participation or, in the investigator's judgment, make the participant inappropriate for the study.

   Prior/Concomitant Therapy:
7. Use of prescription or nonprescription drugs and dietary and herbal supplements within 14 days or 5 half-lives (whichever is longer) prior to the first dose of study intervention. Prior/Concurrent Clinical Study Experience:
8. Previous administration with an investigational drug within 30 days (or as determined by the local requirement) or 5 half-lives preceding the first dose of study intervention used in this study (whichever is longer).

   Diagnostic Assessments:
9. A positive urine drug test.
10. Has participated in, is currently participating in, or is seeking treatment for substance-and/or alcohol-related disorders (excluding nicotine and caffeine).
11. Has a positive alcohol breathalyzer test at screening or upon admission to the study center of Treatment Period. Positive results may be repeated and/or participants re-scheduled at the investigator's discretions.
12. Screening supine BP ≥140 mm Hg (systolic) or ≥90 mm Hg (diastolic), following at least 5 minutes of supine rest. If BP is ≥140 mm Hg (systolic) or ≥90 mm Hg (diastolic), the BP should be repeated 2 more times and the average of the 3 BP values should be used to determine the participant's eligibility. Repeated BP tests should be spaced at least 5 minutes apart.
13. Screening supine 12-lead ECG demonstrating a QTc interval > 450 msec or a QRS interval > 120 msec. If QTc exceeds 450 msec, or QRS exceeds 120 msec, the ECG should be repeated 2 more times and the average of the 3 QTc or QRS values should be used to determine the participant's eligibility.
14. Participants with ANY of the following abnormalities in clinical laboratory tests at screening, as assessed by the study-specific laboratory and confirmed by a single repeat test, if deemed necessary:

    Abnormal platelet count and/or PT/INR; AST or ALT level ≥1.5 × ULN; Total bilirubin level ≥1.5 × ULN; participants with a history of Gilbert's syndrome may have direct bilirubin measured and would be eligible for this study provided the direct bilirubin level is ≤ ULN.

    Other Exclusions:
15. Blood donation (excluding plasma donations) of approximately 1 pint (500 mL) or more within 60 days prior to dosing.
16. History of sensitivity to heparin or heparin-induced thrombocytopenia.
17. Unwilling or unable to comply with the criteria in the Lifestyle Considerations section of this protocol.
18. History of hypersensitivity to naloxone or any of the components in the formulation of the study products.
19. Investigator site staff or Pfizer employees directly involved in the conduct of the study, site staff otherwise supervised by the investigator, and their respective family members.

    -

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 13 (Actual)
Dates: Start 2020-10-06 (Actual); Primary Completion 2021-01-08 (Actual); Study Completion 2021-01-08 (Actual)

PRIMARY OUTCOMES:
Maximum observed plasma naloxone concentration (Cmax) of a single 5 mg IM autoinjector injection compared to a 2 mg IM injection | predose, 2.5, 5, 10, 15, 30, 45, 60, 90, 120, 180, 240, 360, 480, and 1440 minutes after dose
  Comparison of bioavailability
Area under the naloxone concentration versus time curve (AUC) from time zero to the last collection time (AUClast) of a single 5 mg IM autoinjector injection compared to a 2 mg IM injection | predose, 2.5, 5, 10, 15, 30, 45, 60, 90, 120, 180, 240, 360, 480, and 1440 minutes after dose
  Comparison of bioavailability

SECONDARY OUTCOMES:
AUC from time zero to 2.5 minutes (AUC0-2.5) | predose and 2.5 minutes after dose
  Pharmacokinetics all treatment arms
AUC from time zero to 5 minutes (AUC0-5) | predose, 2.5 and 5 minutes after dose
  Pharmacokinetics all treatment arms
AUC from time zero to 15 minutes (AUC0-15) | predose, 2.5, 5, 10 and 15 minutes after dose
  Pharmacokinetics all treatment arms
AUC from time zero to 30 minutes (AUC0-30) | predose, 2.5, 5, 10, 15, and 30 minutes after dose
  Pharmacokinetics all treatment arms
AUC from time zero extrapolated to infinity (AUCinf) [if data permit] | predose, 2.5, 5, 10, 15, 30, 60,90, 120, 180, 240, 360, 480, 1440 minutes after dose
  Pharmacokinetics all treatment arms
Time to maximum observed naloxone plasma concentration (Tmax) [if data permit], | predose, 2.5, 5, 10, 15, 30, 60,90, 120, 180, 240, 360, 480, 1440 minutes after dose
  Pharmacokinetics all treatment arms
Time for naloxone plasma concentration to decrease by one half (t1/2) [if data permit]. | predose, 2.5, 5, 10, 15, 30, 60,90, 120, 180, 240, 360, 480, 1440 minutes after dose
  Pharmacokinetics all treatment arms
Number of participants with a clinically significant change from baseline physical examination | baseline to 28 days after last dose
  Safety and tolerability all treatments
Number of participants with a clinically significant change from baseline vital signs | baseline to 28 days after last dose
  Safety and tolerability all treatments
Number of participants with a clinically significant change from baseline clinical safety laboratory measurements | baseline to 28 days after last dose
  Safety and tolerability all treatment arms
Number of participants with clinically significant AEs from baseline | baseline to 28 days after last dose
  Safety and tolerability all treatment arms

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- New Haven Clinical Research Unit, New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=C2431001